CLINICAL TRIAL: NCT02041195
Title: A Staged, Phase 1b/Phase 2a, Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety and Efficacy of RM-493, a Melanocortin 4 Receptor (MC4R) Agonist in Obese Patients Using a Once or Twice Daily Sub-Cutaneous Injection Formulation
Brief Title: Phase 1b/2a Study to Evaluate Safety and Efficacy of Setmelanotide in Obese Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM-493-009
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Results first posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Overweight and Obesity
Keywords: Overweight
MeSH Terms: conditions — Overweight; Obesity | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Setmelanotide Once Daily (Active Comparator): Once daily in the morning, equivalent placebo in evening.
  Interventions: Drug: Setmelanotide; Drug: Placebo
- Setmelanotide Split Dose (Active Comparator): Split dose, one half in the morning and one half in the evening.
  Interventions: Drug: Setmelanotide
- Placebo (Placebo Comparator): Placebo in the morning, placebo in the evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Setmelanotide
  Other Names: RM-493
  Arms: Setmelanotide Once Daily; Setmelanotide Split Dose
Drug: Placebo
  Arms: Placebo; Setmelanotide Once Daily

SUMMARY:
The purpose of this study is to evaluate the effects of a new daily subcutaneous (SC) injectable formulation of setmelanotide (RM-493) in healthy participants with obesity on mean percent body weight loss and other weight loss parameters, as well as pharmacokinetic (PK) profile. The study is designed to evaluate the efficacy and tolerability of setmelanotide administered once or twice daily. The study drug (setmelanotide and placebo) will be administered in a blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 65 years, inclusive.
* Able to provide voluntary, written informed consent with comprehension of all aspects of the protocol, prior to any study procedures.
* In good general health, without significant medical history, physical examination findings, or clinical laboratory abnormalities.
* Body Mass Index: 30 to 40 Kg/m2.
* Stable body weight by participant report (+/- 5 Kg) during previous 6 months.
* Blood pressure (<140/90 mmHg); may include stable dose (≥ 30 days of use) of up to two anti-hypertensive medications to achieve control and that are intended to remain on a stable dose during the protocol.
* Willingness (during screening) and demonstrated ability (as witnessed in the clinic prior to randomization) to self-administer study medication subcutaneously via a once or twice daily SC injection using a small insulin syringe.
* Willing to maintain a healthy diet and exercise regime throughout study as recommended by counseling at study start.
* Female participants must have negative serum pregnancy test and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method (i.e., sponge), or a double-barrier method of birth control (i.e., condom with spermicide) or abstinence must be used/ practiced throughout the study and for 90 days following the study.
* Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months (and confirmed with a screening FSH level in the post-menopausal lab range), do not require contraception during the study.
* Males with female partners of childbearing potential must agree to a double barrier method if they become sexually active during the study and for 90 days following the study. Male participants must not donate sperm for 90 days following their participation in the study.

Exclusion Criteria:

* Fasting blood glucose > than 140 mg/dL.
* TSH level outside the normal range.
* Creatinine > 1.5 times the upper limit of normal.
* Liver function tests > 2 times the upper limit of normal.
* Active or history of any significant medical condition including renal, hepatic, pulmonary, gastrointestinal, cardiovascular, genitourinary, endocrine, immunologic, metabolic, neurologic or hematological disease.
* Patients with a history of the following:

  1. Uncontrolled hypertension;
  2. Diabetes requiring medical treatment;
  3. Major depressive disorder within the last 2 years;
  4. Any lifetime history of a suicide attempt;
  5. Any suicidal ideation/behavior in the last month;
  6. Other severe psychiatric disorders (e.g. schizophrenia, bipolar disorder, severe eating disorders including bulimia).
* A PHQ-9 score of ≥15.
* Any suicidal ideation of type 4 or 5 on the C-SSRS.
* Prior bariatric surgery.
* History or close family history (parents or siblings) of melanoma.
* Significant dermatologic findings as part of the Screening comprehensive skin evaluation performed by the dermatologist.
* Currently treated with anorectic agents or drugs in last 2 months from screening with anorexia as a frequent side event.
* Taking more than 2 anti-hypertensive medications.
* Acute illness or history of illness, which in the opinion of the Investigator, could pose a threat or harm to the patient or obscure interpretation of laboratory test results or interpretation of study data.
* History of any malignancy, past or present, including skin cancer, multiple severely dysplastic nevi, or nevoid basal cell carcinoma.
* History of HIV infection or Hepatitis B or C.
* History of significant drug hypersensitivity or anaphylaxis.
* History of hypersensitivity to proteins (e.g., allergy shots).
* Any clinically significant abnormalities on screening laboratories as determined by the Investigator.
* Abnormal 12-lead electrocardiogram (ECG) at screening, except minor deviations deemed to be of no clinical significance by the Investigator. QTcF must be < 450 ms.
* Received any experimental drugs or devices or have participated in a clinical study within 30 days prior to dosing.
* Blood donation greater than 500 mL within 60 days prior to screening or intent to donate up to 30 days after Final Study Visit.
* Hospitalization for surgery within the 3 months prior to screening except for minor outpatient procedures, or any planned hospitalizations during the study period.
* Poor venous access or inability to tolerate venipuncture.
* Inability to attend all study visits or comply with protocol requirements including fasting and restrictions on concomitant medication intake.
* Participation in weight loss programs during the study period, including nutritional supplements/ replacements other than as recommended by nutritional counseling provided at study start.
* Use of prescription medications on a regular basis with the following exceptions:

  1. Contraceptives (must be on for ≥3 months);
  2. Hormone replacement therapy (must be on stable dose for ≥3 months);
  3. Antihypertensives (<2 medications on a stable dose for ≥ 30 days);
  4. Statins (dose must be ≤ half the maximum dose; must be on a stable dose ≥3 months);
  5. Thyroxin (stable dose for ≥ 30 days);
  6. The last use of any other prescription medication must have been greater than 5 half-lives for the specific medication or at least 14 days prior to randomization, whichever is longer.
* Women who are pregnant or are breast feeding.
* Previously randomized and dosed in this study or previously exposed to setmelanotide.
* History of alcohol or drug abuse within 5 years of Screening Visit.
* Any other reason, which in the opinion of the Investigator, would confound proper evaluation of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Meeker, MD, Study Chair — Rhythm Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Dallas, Texas
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage A: Setmelanotide 0.75 mg BID: Participants received setmelanotide 0.75 milligrams (mg) by subcutaneous (SC) injection twice daily (BID) for approximately 4 weeks while housed in the Phase 1 unit. During the first 4 weeks, participants were advanced to setmelanotide 2 mg SC BID. Thereafter, participants received setmelanotide 2 mg once daily (QD) by SC injection for the rest of the 12-week study with drug self-administration as outpatients.
- Stage A: Setmelanotide 1.5 mg QD: Participants received setmelanotide 1.5 mg by SC injection QD for approximately 4 weeks while housed in the Phase 1 unit. During the first 4 weeks, participants were advanced to setmelanotide 2 mg once daily. Thereafter, participants received setmelanotide 2 mg once daily by SC injection for the rest of the 12-week study with drug self-administration as outpatients.
- Stage A: Placebo 0.75 mg BID: Participants received placebo matched to setmelanotide by SC injection BID for approximately 4 weeks while housed in the Phase 1 unit. Thereafter, participants received placebo matched to setmelanotide QD by SC injection for the rest of the 12-week study with drug self-administration as outpatients.
- Stage A: Placebo 1.5 mg QD: Participants received placebo matched to setmelanotide by SC injection QD for approximately 4 weeks while housed in the Phase 1 unit. Thereafter, participants received placebo matched to setmelanotide QD by SC injection for the rest of the 12-week study with drug self-administration as outpatients.
- Stage B: Setmelanotide 1.5 mg QD: Participants initially received setmelanotide 1.5 mg QD and then advanced to 2 mg QD for the remainder of the 12-week treatment period. All participants self-administered the study drug.
- Stage B: Placebo 1.5 mg QD; Stage C: Placebo 2 mg QD: Participants received placebo matched to setmelanotide QD for the 12-week treatment period. All participants self-administered the study drug.
- Stage C: Setmelanotide 2 mg QD: Participants received setmelanotide 2 mg QD for the 12-week treatment period. All participants self-administered the study drug.
Period: Overall Study
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD | Stage A: Placebo 0.75 mg BID | Stage A: Placebo 1.5 mg QD | Stage B: Setmelanotide 1.5 mg QD | Stage B: Placebo 1.5 mg QD | Stage C: Setmelanotide 2 mg QD | Stage C: Placebo 2 mg QD
Started | 10 | 9 | 3 | 3 | 11 | 6 | 29 | 28
Completed | 8 | 6 | 3 | 3 | 10 | 6 | 22 | 25
Not Completed | 2 | 3 | 0 | 0 | 1 | 0 | 7 | 3
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Not completed — Unable to comply with study visits | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of study drug and had a post-baseline observation.
Groups:
- Stage A: Setmelanotide 0.75 mg BID: Participants received setmelanotide 0.75 mg by SC injection BID for approximately 4 weeks while housed in the Phase 1 unit. During the first 4 weeks, participants were advanced to setmelanotide 2 mg SC BID. Thereafter, participants received setmelanotide 2 mg QD by SC injection for the rest of the 12-week study with drug self-administration as outpatients.
- Total: Total of all reporting groups
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD | Stage A: Placebo 0.75 mg BID | Stage A: Placebo 1.5 mg QD | Stage B: Setmelanotide 1.5 mg QD | Stage B: Placebo 1.5 mg QD | Stage C: Setmelanotide 2 mg QD | Stage C: Placebo 2 mg QD | Total
Number analyzed (Participants) | 10 | 9 | 3 | 3 | 11 | 6 | 29 | 28 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 3 | 3 | 11 | 6 | 29 | 28 | 99
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 1 | 1 | 5 | 4 | 21 | 18 | 59
  Male | 4 | 6 | 2 | 2 | 6 | 2 | 8 | 10 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 2 | 0 | 1 | 2 | 3 | 3 | 17
  Not Hispanic or Latino | 9 | 4 | 1 | 3 | 10 | 4 | 26 | 25 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Black or African American | 8 | 4 | 1 | 2 | 5 | 4 | 11 | 9 | 44
  White | 2 | 4 | 1 | 1 | 6 | 2 | 13 | 17 | 46
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 3 | 3 | 11 | 6 | 29 | 28 | 99

OUTCOME MEASURES:

1. Primary Outcome: Body Weight - Stage A
Time Frame: Baseline
Population: Full Analysis Set (FAS) included all participants with a baseline and at least one post-dose efficacy observation. Data from 2 placebo groups were combined for the efficacy analysis.
Measure: Mean (Standard Error); unit: Kilograms (kg)
Groups:
- Stage A: Placebo: Participants received placebo matched to setmelanotide by SC injection QD or BID for approximately 4 weeks while housed in the Phase 1 unit. Thereafter, participants received placebo matched to setmelanotide QD by SC injection for the rest of the 12-week study with drug self-administration as outpatients.
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD | Stage A: Placebo
Number analyzed (Participants) | 10 | 9 | 6
Kilograms (kg) | 101.7 (5.09) | 101.7 (4.24) | 94.5 (3.85)

2. Primary Outcome: Percent Change From Baseline in Body Weight at Week 12 - Stage A
Time Frame: Baseline, Week 12
Population: Participants in the FAS with available data were analyzed. Data from 2 placebo groups were combined for the efficacy analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD | Stage A: Placebo
Number analyzed (Participants) | 8 | 6 | 6
percent change | -1.38 [-3.27 to 0.52] | -0.74 [-2.77 to 1.28] | 2.89 [0.53 to 5.25]
Statistical Analysis 1: Comparison: Stage A: Setmelanotide 0.75 mg BID vs Stage A: Placebo; Test type: Other; p = 0.004, Longitudinal mixed analysis of variance — One sided p-value; Least Squares (LS) Mean Difference = -4.26, 90% CI 2-sided [-6.81 to -1.72] — A longitudinal mixed analysis of variance model with fixed effects for treatment, timepoint, treatment-by-timepoint, baseline weight as covariate, and participant as random effect was used
Statistical Analysis 2: Comparison: Stage A: Setmelanotide 1.5 mg QD vs Stage A: Placebo; Test type: Other; p = 0.012, Longitudinal mixed analysis of variance; One-sided p-value; LS Mean difference = -3.63, 90% CI 2-sided [-6.23 to -1.03] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Body Weight - Stage B
Time Frame: Baseline
Population: Participants in the FAS were analyzed.
Measure: Mean (Standard Error); unit: kg
Arm/Group | Stage B: Setmelanotide 1.5 mg QD | Stage B: Placebo 1.5 mg QD
Number analyzed (Participants) | 11 | 6
kg | 99.4 (3.51) | 93.3 (2.92)

4. Primary Outcome: Percent Change From Baseline in Body Weight at Week 12 - Stage B
Time Frame: Baseline, Week 12
Population: Participants in the FAS with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Stage B: Setmelanotide 1.5 mg QD | Stage B: Placebo 1.5 mg QD
Number analyzed (Participants) | 10 | 5
percent change | -1.29 [-2.47 to -0.11] | 2.28 [0.68 to 3.88]
Statistical Analysis 1: Comparison: Stage B: Setmelanotide 1.5 mg QD vs Stage B: Placebo 1.5 mg QD; Test type: Other; p < 0.001, Longitudinal mixed analysis of variance — One sided p-value; LS Mean Difference = -3.57, 90% CI 2-sided [-5.24 to -1.89] — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Body Weight - Stage C
Time Frame: Baseline
Population: Participants in the FAS were analyzed.
Measure: Mean (Standard Error); unit: Kg
Arm/Group | Stage C: Setmelanotide 2 mg QD | Stage C: Placebo 2 mg QD
Number analyzed (Participants) | 29 | 28
Kg | 98.5 (1.87) | 98.7 (2.44)

6. Primary Outcome: Percent Change From Baseline in Body Weight at Week 12 - Stage C
Time Frame: Baseline, Week 12
Population: Participants in the FAS with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Stage C: Setmelanotide 2 mg QD | Stage C: Placebo 2 mg QD
Number analyzed (Participants) | 22 | 25
percent change | -2.28 [-3.32 to -1.25] | -0.06 [-1.08 to 0.95]
Statistical Analysis 1: Comparison: Stage C: Setmelanotide 2 mg QD vs Stage C: Placebo 2 mg QD; Test type: Other; p = 0.002, Longitudinal mixed analysis of variance; LS Mean Difference = -2.22, 90% CI 2-sided [-3.44 to -1.00] — [estimate comment as in outcome 2, analysis 1]

7. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) - Stage A
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. AEs that occurred after the start of study drug administration were considered TEAEs.
Time Frame: From first dose up to Day 114
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD | Stage A: Placebo 0.75 mg BID | Stage A: Placebo 1.5 mg QD
Number analyzed (Participants) | 10 | 9 | 3 | 3
Participants | 10 | 8 | 2 | 3

8. Primary Outcome: Number of Participants With TEAEs - Stage B
Description: An AE was any untoward medical occurrence in a clinical trial participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. AEs that occurred after the start of study drug administration were considered TEAEs.
Time Frame: From first dose up to Day 114
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage B: Setmelanotide 1.5 mg QD | Stage B: Placebo 1.5 mg QD
Number analyzed (Participants) | 11 | 6
Participants | 9 | 3

9. Primary Outcome: Number of Participants With TEAEs - Stage C
Description: as for outcome 8
Time Frame: From first dose up to Day 114
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Stage C: Setmelanotide 2 mg QD | Stage C: Placebo 2 mg QD
Number analyzed (Participants) | 29 | 28
Participants | 29 | 21

10. Secondary Outcome: Mean Setmelanotide Concentrations During a 24-Hour Steady State Interval on Day 8 - Stage A
Time Frame: Predose (0 hours) and at 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 22, and 24 hours after dosing on Day 8
Population: Participants in the Pharmacokinetic (PK) Evaluable Population (included all participants who received at least 1 dose of study drug, had a post-baseline observation and had evaluable plasma concentration-time profiles for setmelanotide) with available data were analyzed
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD
Number analyzed (Participants) | 9 | 9
nanograms per milliliter (ng/mL)
  Predose (0 hours) | 7.24 (2.52) | 3.54 (0.949)
  1 hour postdose | 9.18 (3.04) | 8.51 (3.07)
  2 hours postdose | 10.8 (3.93) | 13.0 (5.75)
  4 hours postdose | 13.9 (5.05) | 18.0 (6.26)
  6 hours postdose | 11.8 (5.02) | 20.6 (5.27)
  8 hours postdose | 9.86 (3.66) | 19.8 (3.19)
  10 hours postdose | 7.48 (3.18) | 15.5 (2.46)
  12 hours postdose | 6.02 (2.49) | 11.1 (1.63)
  14 hours postdose: number analyzed (Participants) | 8 | 9
  14 hours postdose | 10.6 (5.65) | 9.15 (1.29)
  16 hours postdose | 13.6 (6.96) | 7.32 (1.15)
  20 hours postdose | 9.26 (3.86) | 5.23 (0.991)
  22 hours postdose | 7.43 (3.32) | 4.41 (0.945)
  24 hours postdose | 5.74 (2.72) | 3.58 (0.900)

11. Secondary Outcome: Mean Setmelanotide Concentrations During a 24-Hour Steady State Interval on Day 8 - Stage C
Time Frame: Predose (0 hours) and at 1, 2, 4, 6, 8, 10, 12, 14 and 24 hours after dosing on Day 8
Population: The PK Evaluable Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage C: Setmelanotide 2 mg QD
Number analyzed (Participants) | 12
ng/mL
  Predose (0 hours) | 5.03 (1.84)
  1 hour postdose | 12.3 (3.99)
  2 hours postdose | 18.1 (6.23)
  4 hours postdose | 24.2 (8.19)
  6 hours postdose | 26.5 (7.32)
  8 hours postdose | 24.0 (5.88)
  10 hours postdose | 18.1 (3.76)
  12 hours postdose | 13.9 (3.35)
  14 hours postdose | 11.2 (2.47)
  24 hours postdose | 4.74 (1.66)

12. Secondary Outcome: Change From Baseline in Ambulatory Blood Pressure Monitoring (ABPM) Parameters During 24-Hour Interval Between Days 8 and 15 - Stage A
Description: The 24-hour ABPM parameters were obtained twice once at Baseline and once during 24-hour interval between Days 8 and 15 for all participants in Stage A. Change from Baseline in ABPM parameters (systolic blood pressure [SBP], diastolic blood pressure [DBP], pulse pressure, mean arterial pressure [MAP]) during 24-hour interval between Days 8 and 15 is presented.
Time Frame: Baseline and for one 24-hour interval between Days 8 or 15
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD | Stage A: Placebo 0.75 mg BID | Stage A: Placebo 1.5 mg QD
Number analyzed (Participants) | 10 | 8 | 3 | 3
millimeters of mercury (mmHg)
  Baseline: SBP | 121.09 (7.18) | 119.89 (10.36) | 115.31 (3.81) | 117.01 (10.09)
  Change at 24-hour interval between Days 8 and 15: SBP: number analyzed (Participants) | 9 | 8 | 3 | 3
  Change at 24-hour interval between Days 8 and 15: SBP | -4.08 (6.55) | -2.23 (3.95) | -0.67 (4.61) | -1.08 (2.90)
  Baseline: DBP | 71.02 (5.03) | 73.09 (9.22) | 70.48 (1.35) | 71.08 (8.81)
  Change at 24-hour interval between Days 8 and 15: DBP: number analyzed (Participants) | 9 | 8 | 3 | 3
  Change at 24-hour interval between Days 8 and 15: DBP | -2.13 (3.93) | -1.55 (2.63) | 0.58 (3.42) | -1.90 (2.47)
  Baseline: Pulse pressure | 50.07 (4.77) | 46.79 (5.31) | 44.83 (3.20) | 45.93 (2.07)
  Change at 24-hour interval between Days 8 and 15: Pulse pressure: number analyzed (Participants) | 9 | 8 | 3 | 3
  Change at 24-hour interval between Days 8 and 15: Pulse pressure | -1.94 (3.89) | -0.68 (2.32) | -1.25 (3.10) | 0.82 (0.77)
  Baseline: MAP | 88.27 (5.50) | 89.05 (8.69) | 85.45 (2.05) | 86.85 (8.34)
  Change at 24-hour interval between Days 8 and 15: MAP: number analyzed (Participants) | 9 | 8 | 3 | 3
  Change at 24-hour interval between Days 8 and 15: MAP | -2.73 (4.42) | -1.98 (2.81) | 0.44 (3.46) | -1.63 (2.67)

13. Secondary Outcome: Change From Baseline in ABPM Parameters During 24-Hour Interval Between Days 8 and 15 - Stage C
Description: The 24-hour ABPM parameters were obtained twice once at Baseline and once during 24-hour interval between Days 8 and 15 for a subset of participants in Stage C. Change from Baseline in ABPM parameters (SBP, DBP, pulse pressure, MAP) during 24-hour interval between Days 8 and 15 is presented.
Time Frame: Baseline and for one 24-hour interval between Days 8 or 15
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Stage C: Setmelanotide 2 mg QD | Stage C: Placebo 2 mg QD
Number analyzed (Participants) | 17 | 16
mmHg
  Baseline: SBP | 117.57 (9.99) | 117.51 (8.05)
  Change at 24-hour interval between Days 8 and 15: SBP: number analyzed (Participants) | 17 | 15
  Change at 24-hour interval between Days 8 and 15: SBP | 1.63 (6.83) | 1.22 (6.28)
  Baseline: DBP | 68.90 (7.57) | 69.92 (5.96)
  Change at 24-hour interval between Days 8 and 15: DBP: number analyzed (Participants) | 17 | 15
  Change at 24-hour interval between Days 8 and 15: DBP | 1.77 (4.83) | 0.83 (4.32)
  Baseline: Pulse pressure | 48.67 (7.46) | 47.59 (7.58)
  Change at 24-hour interval between Days 8 and 15: Pulse pressure: number analyzed (Participants) | 17 | 15
  Change at 24-hour interval between Days 8 and 15: Pulse pressure | -0.14 (3.39) | 0.38 (2.70)
  Baseline: MAP | 85.97 (7.33) | 86.30 (5.23)
  Change at 24-hour interval between Days 8 and 15: MAP: number analyzed (Participants) | 17 | 15
  Change at 24-hour interval between Days 8 and 15: MAP | 1.21 (5.35) | 0.68 (4.56)

14. Secondary Outcome: Change From Baseline in Heart Rate Using ABPM During 24-Hour Interval Between Days 8 and 15 - Stage A
Description: The 24-hour ABPM parameters were obtained twice once at Baseline and once during 24-hour interval between Days 8 and 15 for all participants in Stage A. Change from Baseline in heart rate during 24-hour interval between Days 8 and 15 is presented.
Time Frame: Baseline and for one 24-hour interval between Days 8 and 15
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD | Stage A: Placebo 0.75 mg BID | Stage A: Placebo 1.5 mg QD
Number analyzed (Participants) | 10 | 8 | 3 | 3
beats per minute (bpm)
  Baseline | 79.28 (7.05) | 77.55 (8.21) | 72.92 (6.80) | 68.10 (6.48)
  Change at 24-hour interval between Days 8 and 15: number analyzed (Participants) | 9 | 8 | 3 | 3
  Change at 24-hour interval between Days 8 and 15 | -0.90 (3.87) | -2.70 (5.38) | -5.75 (7.72) | 1.35 (7.70)

15. Secondary Outcome: Change From Baseline in Heart Rate Using ABPM During 24-Hour Interval Between Days 8 and 15 - Stage C
Description: The 24-hour ABPM parameters were obtained twice once at Baseline and once during 24-hour interval between Days 8 and 15 for a subset of participants in Stage C. Change from Baseline in heart rate during 24-hour interval between Days 8 and 15 is presented.
Time Frame: Baseline and for one 24-hour interval between Days 8 and 15
Population: Participants in the FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Stage C: Setmelanotide 2 mg QD | Stage C: Placebo 2 mg QD
Number analyzed (Participants) | 17 | 16
bpm
  Baseline | 80.77 (9.03) | 73.01 (10.65)
  Change at 24-hour interval between Days 8 and 15: number analyzed (Participants) | 17 | 15
  Change at 24-hour interval between Days 8 and 15 | -0.95 (9.78) | 0.98 (4.21)

ADVERSE EVENTS:
Time Frame: From first dose up to Day 114
Description: Safety Population
Arm/Group | Stage A: Setmelanotide 0.75 mg BID | Stage A: Setmelanotide 1.5 mg QD | Stage A: Placebo 0.75 mg BID | Stage A: Placebo 1.5 mg QD | Stage B: Setmelanotide 1.5 mg QD | Stage B: Placebo 1.5 mg QD | Stage C: Setmelanotide 2 mg QD | Stage C: Placebo 2 mg QD
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/3 | 0/3 | 0/11 | 0/6 | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/3 | 0/3 | 0/11 | 0/6 | 1/29 | 1/28
Other Adverse Events (participants affected / at risk) | 10/10 | 8/9 | 2/3 | 3/3 | 9/11 | 3/6 | 29/29 | 21/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage A: Setmelanotide 0.75 mg BID (N=10) | Stage A: Setmelanotide 1.5 mg QD (N=9) | Stage A: Placebo 0.75 mg BID (N=3) | Stage A: Placebo 1.5 mg QD (N=3) | Stage B: Setmelanotide 1.5 mg QD (N=11) | Stage B: Placebo 1.5 mg QD (N=6) | Stage C: Setmelanotide 2 mg QD (N=29) | Stage C: Placebo 2 mg QD (N=28)
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage A: Setmelanotide 0.75 mg BID (N=10) | Stage A: Setmelanotide 1.5 mg QD (N=9) | Stage A: Placebo 0.75 mg BID (N=3) | Stage A: Placebo 1.5 mg QD (N=3) | Stage B: Setmelanotide 1.5 mg QD (N=11) | Stage B: Placebo 1.5 mg QD (N=6) | Stage C: Setmelanotide 2 mg QD (N=29) | Stage C: Placebo 2 mg QD (N=28)
Nausea (Gastrointestinal disorders) | 3 | 6 | 0 | 1 | 6 | 1 | 17 | 3
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 3 | 1 | 10 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3 | 1 | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 | 6 | 1 | 0 | 8 | 0 | 26 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 2 | 0
Injection site erythema (General disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 7 | 4
Fatigue (General disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 10 | 2
Injection site pain (General disorders) | 1 | 3 | 0 | 0 | 1 | 1 | 2 | 2
Pain (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 5 | 4 | 0 | 0 | 4 | 2 | 16 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 2 | 0 | 1 | 2
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 3 | 0 | 0 | 3 | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 10 | 4
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 4 | 2 | 0 | 0 | 2 | 0 | 5 | 0
Injection site swelling (General disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Injection site induration (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injury associated with device (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site scar (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site warmth (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine spasm (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulva cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginismus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scleral discolouration (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye colour change (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 6
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 3 | 0 | 10 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in sexual arousal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Logorrhoea (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No